CLINICAL TRIAL: NCT02948127
Title: Phase I Placebo-Controlled Study of the Infectivity, Safety and Immunogenicity of a Single Dose of a Recombinant Live-attenuated Respiratory Syncytial Virus Vaccine, LID cp ΔM2-2, Lot RSV#009B, Delivered as Nose Drops to RSV-Seronegative Infants and Children 6 to 24 Months of Age
Brief Title: Infectivity, Safety and Immunogenicity of a Recombinant Live-Attenuated Respiratory Syncytial Virus Vaccine (RSV LID cp ΔM2-2) in RSV-Seronegative Infants and Children 6 to 24 Months of Age
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CIR 312
Record Dates: First submitted 2016-10-25; First posted 2016-10-28 (Estimated); Last update posted 2018-08-17 (Actual); Status verified 2018-08

CONDITIONS: Respiratory Syncytial Virus Infections
MeSH Terms: conditions — Respiratory Syncytial Virus Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- RSV LID cp ΔM2-2 Vaccine (Experimental): Participants will receive a single dose of the RSV LID cp ΔM2-2 vaccine at study entry (Day 0).
  Interventions: Biological: RSV LID cp ΔM2-2 Vaccine
- Placebo (Placebo Comparator): Participants will receive a single dose of placebo at study entry (Day 0).
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: RSV LID cp ΔM2-2 Vaccine — 10^5 plaque-forming units (PFUs); administered as nose drops
  Arms: RSV LID cp ΔM2-2 Vaccine
Biological: Placebo — Administered as nose drops
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, infectivity, and immunogenicity of a single dose of a recombinant live-attenuated respiratory syncytial virus (RSV) vaccine in RSV-seronegative infants and children 6 to 24 months of age.

This study is a companion study to IMPAACT 2012.

DETAILED DESCRIPTION:
Human respiratory syncytial virus (RSV) is the most common viral cause of serious acute lower respiratory illness (LRI) in infants and children under 5 years of age worldwide. This study will evaluate the safety, infectivity, and immunogenicity of a single dose of RSV LID cp ΔM2-2, a recombinant live-attenuated RSV vaccine, in RSV-seronegative infants and children 6 to 24 months of age.

Participants will be randomly assigned to receive a single dose of the RSV LID cp ΔM2-2 vaccine or placebo at study entry (Day 0).

Participants will be enrolled in the study between April 1 and October 31 (outside of RSV season) and will remain on study until they complete the post-RSV season visit between April 1 and April 30 in the calendar year following enrollment. Participants' total study duration will be between 6 and 13 months, depending on when they enroll in the study. Participants will be evaluated in study visits that may include physical examinations, blood collection, and nasal washes. Additionally, participants' parents or guardians will be contacted by study staff at various times during the study to monitor participants' health.

ELIGIBILITY:
Inclusion Criteria:

* Greater than or equal to 6 months (greater than or equal to 180 days) of age at the time of screening and less than 25 months (less than 750 days) of age
* Participant is in good health based on review of the medical record, history, and physical examination, without evidence of chronic disease
* Parents/guardians are willing and able to provide written informed consent
* Seronegative for RSV antibody, defined as a serum RSV-neutralizing antibody titer less than 1:40 at screening from a sample collected no more than 42 days prior to inoculation
* Is growing at a normal velocity for age as demonstrated on a standard growth chart AND

  * If less than 1 year of age: has a current height and weight above the 5th percentile
  * If 1 year of age or older: has a current height and weight above the 3rd percentile for age
* Participant has received routine immunizations appropriate for age (as per Center for Disease Control Advisory Committee on Immunization Practices [ACIP])
* Participant is expected to be available for the duration of the study

Exclusion Criteria:

* Known or suspected HIV infection or impairment of immunological functions
* Receipt of immunosuppressive therapy, including any systemic, including either nasal or inhaled, corticosteroids within 28 days of enrollment. Note: Cutaneous (topical) steroid treatment is not an exclusion.
* Bone marrow/solid organ transplant recipient
* Major congenital malformations (such as congenital cleft palate) or cytogenetic abnormalities
* Previous receipt of a licensed or investigational RSV vaccine or receipt of placebo in any IMPAACT RSV study or previous receipt of or planned administration of any anti-RSV product (such as ribavirin or RSV Ig or RSV mAb)
* Previous anaphylactic reaction
* Previous vaccine-associated adverse reaction that was Grade 3 or above
* Known hypersensitivity to any study product component
* Heart disease. Note: Participants with cardiac abnormalities documented to be clinically insignificant and requiring no treatment may be enrolled
* Lung disease, including any history of reactive airway disease or medically documented wheezing
* Member of a household that contains, or will contain, an infant who is less than 6 months of age at the enrollment date through Day 28
* Member of a household that contains another child who is, or is scheduled to be, enrolled in CIR 311, 312 or 313 AND there has been or will be an overlap in residency during that other child's participation in the study's Acute Phase (Days 0 to 28)
* Member of a household that contains an immunocompromised individual, including but not limited to:

  * a person who is HIV infected
  * a person who has received chemotherapy within the 12 months prior to enrollment
  * a person receiving immunosuppressant agents
  * a person living with a solid organ or bone marrow transplant
* Attends a daycare facility and shares a room with infants less than 6 months of age, and parent/guardian is unable or unwilling to suspend daycare for 28 days following inoculation
* Any of the following events at the time of enrollment:

  * fever (temporal or rectal temperature of greater than or equal to 100.4°F), or
  * upper respiratory signs or symptoms (rhinorrhea, cough, or pharyngitis) or
  * nasal congestion significant enough to interfere with successful inoculation, or
  * otitis media
* Receipt of the following prior to enrollment:

  * any killed vaccine or live-attenuated rotavirus vaccine within the 14 days prior, or
  * any live vaccine, other than rotavirus vaccine, within the 28 days prior, or
  * another investigational vaccine or investigational drug within 28 days prior
* Scheduled administration of the following after planned inoculation:

  * killed vaccine or live-attenuated rotavirus vaccine within the 14 days after, or
  * any live vaccine other than rotavirus in the 28 days after, or
  * another investigational vaccine or investigational drug in the 56 days after
* Receipt of immunoglobulin, any antibody products, or any blood products within the past 6 months
* Receipt of any of the following medications within 3 days of study enrollment:

  * systemic antibacterial, antiviral, antifungal, anti-parasitic, or antituberculous agents, whether for treatment or prophylaxis, or
  * intranasal medications, or
  * other prescription medication except as listed below
* Receipt of salicylate (aspirin) or salicylate-containing products within the past 28 days
* Born at less than 34 weeks gestation
* Born at less than 37 weeks gestation and less than 1 year of age at the time of enrollment
* Suspected or documented developmental disorder, delay, or other developmental problem
* Previous receipt of supplemental oxygen therapy in a home setting

Ages: 6 Months to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 8 (Actual)
Dates: Start 2016-09; Primary Completion 2017-04-30 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Grades of study product-related solicited adverse events (AEs) | Measured through Day 28
Grades of study product-related unsolicited AEs | Measured through Day 28
Grades of study product-related serious adverse events (SAEs) | Measured through Day 56
Number of participants with infection with vaccine virus | Measured through Day 56
  Defined as 1) vaccine virus identified in a nasal wash from Study Day 0-28 (a binary outcome based on nasal washes done throughout the study period; Day 0 nasal wash will be counted as baseline) or 2) greater than or equal to 4-fold rise in RSV neutralizing antibody titer from Study Day 0-56
Peak titer of vaccine virus shed | Measured through Day 28
Duration of vaccine virus shedding in nasal washes measured by culture | Measured through Day 28
Duration of vaccine virus shedding in nasal washes measured by RT-PCR | Measured through Day 28
Frequency of a greater than or equal to 4-fold rise in RSV-neutralizing antibody titer | Measured through Day 56
Antibody responses to RSV F glycoprotein as assessed by enzyme-linked immunosorbent assay (ELISA) | Measured through Day 56

SECONDARY OUTCOMES:
Frequency of symptomatic, medically attended respiratory and febrile illness in the vaccine and placebo recipients who experience natural infection with wild-type RSV during the subsequent RSV season | Measured through participant's last study visit, up to a total of 6 to 12 months after study entry depending on when participants enroll in the study
  Will be measured through the subsequent RSV season (November 1 in the calendar year of study entry to March 31 in the calendar year following study entry)
Measurement of antibody responses in the vaccine and placebo recipients who experience natural infection with wt RSV during the subsequent RSV season | Measured at participant's last study visit, up to a total of 6 to 13 months after study entry depending on when participants enroll in the study
  Will be measured at the post-RSV season visit (between April 1 and April 30 in the calendar year following study entry)
Frequency of B cell responses to vaccine | Measured through participant's last study visit, up to a total of 6 to 13 months after study entry depending on when participants enroll in the study
  Will be measured at the post-RSV season visit (between April 1 and April 30 in the calendar year following study entry)

CONTACTS AND LOCATIONS:
Overall Officials: Ruth Karron, MD, Principal Investigator — Center for Immunization Research (CIR), Johns Hopkins Bloomberg School of Public Health (JHSPH)
Locations (3):
- United States (3):
  - Center for Immunization Research, Johns Hopkins Bloomberg School of Public Health, Baltimore, Maryland
  - Center for Immunization Research East, Johns Hopkins Bayview Medical Center Campus, Baltimore, Maryland
  - Center for Immunization Research South, Laurel, Maryland

REFERENCES:
- [Derived] Cunningham CK, Karron R, Muresan P, McFarland EJ, Perlowski C, Libous J, Thumar B, Gnanashanmugam D, Moye J Jr, Schappell E, Barr E, Rexroad V, Aziz M, Deville J, Rutstein R, Yang L, Luongo C, Collins P, Buchholz U; International Maternal Pediatric Adolescent AIDS Clinical Trials (IMPAACT) 2012 Study Team. Live-Attenuated Respiratory Syncytial Virus Vaccine With Deletion of RNA Synthesis Regulatory Protein M2-2 and Cold Passage Mutations Is Overattenuated. Open Forum Infect Dis. 2019 May 6;6(6):ofz212. doi: 10.1093/ofid/ofz212. eCollection 2019 Jun. PMID 31211158